CLINICAL TRIAL: NCT03044327
Title: Development of Novel Non-invasive Inflammometry Following LPS Challenge in Healthy Volunteers
Brief Title: Development of Novel Non-invasive Inflammometry Following Lipopolysaccharide, Endotoxin (LPS) Challenge in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Hohlfeld, Division Director Airway Research, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-03 DONNER
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LPS challenge (Other): LPS inhalation and bronchial instillation
  Interventions: Procedure: LPS challenge

INTERVENTIONS:
Procedure: LPS challenge — LPS inhalation and bronchial instillation

SUMMARY:
The aim of this study is to further profile and develop the Lipopolysaccharide, endotoxin (LPS) challenge models (both by instillation and inhalation) by investigating the utility of various non-invasive monitoring methods.

DETAILED DESCRIPTION:
The hypothesis of the project is that local inflammatory changes in the lung induced by LPS can be captured by gas-enhanced Magnetic resonance imaging (MRI) and analysis of exhaled breath. While MRI is able to provide localized information on inflammatory processes, exhaled breath analysis can capture integral information over time. Assuming that these novel techniques correlate with cellular measures of inflammation, repetitive measurements to investigate onset and duration of action of investigational new drugs will be made possible.

The evaluation whether LPS induced changes in the lung can be captured and monitored by MRI will be performed by correlation of multiple endpoints describing the cellular composition of the airways with variables derived from MRI and breath analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy subjects, aged 18-65 years. Women will be considered for inclusion if they are:

Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).

Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).

* Normal lung function with FEV1 predicted ≥ 80%
* Nonsmokers with a history of less than 1 pack year having been nonsmokers for at least the last five years
* Able and willing to give written informed consent

Exclusion Criteria:

* • Past or present disease, which as judged by the investigator, may affect the outcome of the study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis)

  * Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements
  * Clinically relevant history of allergy as judged by the investigator
  * Patient unable to undergo MRI (e.g. due to claustrophobia, cardiac pacemaker, hypersensitivity to MR i.v. contrast imaging agents)
  * Infections of the lower respiratory tract within 4 weeks before visit 1, visit 2, or visit 3. These patients can be rescreened starting from visit 1.
  * Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs or ECG at Visit 1, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subject's ability to participate in the study
  * Elevated IgE
  * Intake of systemic or inhaled steroids in the previous 4 weeks before visit 1, visit 2, or visit 3
  * History of drug or alcohol abuse
  * Risk of non-compliance with study procedures
  * Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the number of total cells in bronchoalveolar lavage | change from baseline to 6 hours and 24 hours post LPS

SECONDARY OUTCOMES:
The regional change in xenon uptake in dissolved-phase MRI | change from baseline to 6 hours and 24 hours post LPS
The regional change in oxygen transfer function assessed by MRI | change from baseline to 6 hours and 24 hours post LPS
The change of the number of exhaled particles | change from baseline to 6 hours and 24 hours post LPS

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Principal Investigator — Fraunhofer-Institute of Toxicology and Experimental Medicine
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsson P, Holz O, Koster G, Postle A, Olin AC, Hohlfeld JM. Exhaled breath particles as a novel tool to study lipid composition of epithelial lining fluid from the distal lung. BMC Pulm Med. 2023 Nov 3;23(1):423. doi: 10.1186/s12890-023-02718-8. PMID 37924084
- [Derived] Holz O, Muller M, Carstensen S, Olin AC, Hohlfeld JM. Inflammatory cytokines can be monitored in exhaled breath particles following segmental and inhalation endotoxin challenge in healthy volunteers. Sci Rep. 2022 Apr 4;12(1):5620. doi: 10.1038/s41598-022-09399-z. PMID 35379863